CLINICAL TRIAL: NCT06652256
Title: Fatigue in Systemic Lupus Erythematosus: Which Variables Play a Role?
Brief Title: Fatigue in Systemic Lupus Erythematosus
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Zülal TATAR, Research Assitant, Pamukkale University
Other Study IDs: Fatigue
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Fatigue; Systemic Lupus Erthematosus
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to investigate the effects of biopsychosocial status, quality of life, functional status and hematological markers on fatigue in individuals with SLE.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with SLE according to the 2019 ACR/EULAR diagnostic criteria
* Being 18 years of age or older

Exclusion Criteria:

* Not being able to speak or understand Turkish fluently
* Having a psychiatric illness that will affect cooperation
* Heart failure or lung pathology that will affect daily life activities
* Additional autoimmune disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include individuals aged 18 and older who are receiving treatment for SLE at a university hospital in Turkey, and meet the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Fatigue Assesment Scale | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  It is a scale consisting 10 items. The maximum score is 50. High score indicates high fatigue.
FACIT Fatigue Scale | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  It is scale consisting 13 items. Scores range from 0-52. High score indicates low fatigue

SECONDARY OUTCOMES:
Cognitive Exercise Therapy Approach-Biopsychosocial Questionnaire (BETY-BQ) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  It is a scale consist of 30 items. Scores range from 0-120. Higher scores indicate worse biopsychosocial status.
Short Form 36 (SF-36) Health Survey | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  The SF-36 consists of two dimensions, generating a profile of health-related quality of life.These dimensions are: physical health and mental health. Higher scores indicate better health.
HEALTH ASSESSMENT QUESTIONNAIRE (HAQ) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  The scale consists of 20 questions and includes 8 activities. The total score is obtained by summing the points earned from 8 activities and then dividing that sum by 8. Higher scores indicate worse functional status
Routine blood test results | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Participants' routine blood test results such as neutrophil (NEU (K/uL)) , monocyte (MONO (K/uL)), eosinophil (EO (K/uL)), leukocyte (WBC (K/uL)), lymphocyte (LYM (K/uL)), platelet (PLT (K/uL)) will be recorded.
Routine Blood Test Results | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Participants' routine blood test results such as calcium (Ca (mg/dL)), creatinine (mg/dL), c-reactive protein (CRP (mg/L)), uric acid (mg/dL) will be recorded.
Routine Blood Test Results | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  The participants' rutin blood test such as aspartate aminotransferase (AST IU/L), alanine aminotransferase (ALT IU/L) will be recorded.
Hematological indices | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Neutrophil/lymphocyte (NLR), monocyte/lymphocyte (MLR), platelet/lymphocyte (PLR), platelet*neutrophil/lymphocyte (systemic inflammatory index), monocyte/platelet (MTO), neutrophil*monocyte/lymphocyte (systemic inflammatory response index), neutrophil*monocyte*platelet/lymphocyte (systemic inflammation aggregate index) obtained from complete blood counts will be calculated and recorded.
Routine Blood Test Results | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Procolcytonin (PCT (%)), erythrocyte distribution width (RDW (%)), platelet distribution width (PDW (%)) levels will be recorded.
Routine Blood Test Results | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Erythrocyte distribution width standard deviation (RDW-SD (fL)) will be recorded.
Routine Blood Test Results | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  C3 complement (g/L) and C4 complement (g/L) levels will be recorded.
Routine Blood Test Results | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Blood urea nitrogen (BUN (mg/dL)) levels will be recorded.
Routine Blood Test Results | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Sedimentation (mm/h) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)